CLINICAL TRIAL: NCT06084884
Title: A Phase I/II Open-Label Study to Evaluate the Safety, Cellular Kinetics and Efficacy of AZD5851, a Chimeric Antigen Receptor T-Cell (CAR-T) Therapy Directed Against GPC3 in Adult Participants With Advanced/Recurrent Hepatocellular Carcinoma: ATHENA
Brief Title: A Phase I/II Study to Evaluate AZD5851 in GPC3+ Advanced/Recurrent Hepatocellular Carcinoma
Acronym: ATHENA
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D7670C00001
Record Dates: First submitted 2023-10-03; First posted 2023-10-16 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Liver Cancer; Liver Neoplasm; advanced HCC; HCC; Metastatic Liver Cancer; CAR-T; CART; AZD5851; T-cell; Cell Therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Cell- and Tissue-Based Therapy

STUDY DESIGN:
Masking Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AZD5851 (Experimental): Subjects will receive AZD5851 following 3 consecutive doses of lymphodepleting chemotherapy (fludarabine and cyclophosphamide).
  Interventions: Biological: AZD5851

INTERVENTIONS:
Biological: AZD5851 — Subjects will undergo leukapheresis to isolate peripheral blood mononuclear cells (PBMCs) to produce AZD5851.
  During AZD5851 production, subjects may receive bridging therapy for disease control. Upon successful generation of AZD5851 product, subjects will receive treatment with AZD5851 therapy.
  Study treatment will include lymphodepleting chemotherapy followed by one dose of AZD5851 administered by intravenous (IV) infusion.
  Other Names: Cell Therapy

SUMMARY:
A Phase I/II study to evaluate AZD5851 in patients with GPC3+ advanced/recurrent hepatocellular carcinoma.

DETAILED DESCRIPTION:
This first-time in human, single-arm, open-label multicentre Phase I/II study will evaluate the safety, tolerability, antitumour activity, cellular kinetics, pharmacodynamics, and immunogenicity of AZD5851 in adult participants with GPC3+ advanced/recurrent HCC, where at least one line of prior therapy has failed/or was intolerable, or participant/investigator decision.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 18 years or older and has voluntarily agreed to participate by giving written informed consent.
2. Participants with confirmed advanced/recurrent or metastatic and/or unresectable HCC based on histopathological findings
3. Completed or were unable to tolerate at least one prior line of standard systemic therapy for HCC and/or participant/investigator decision.
4. GPC3-positive tumour as determined by a central laboratory using an analytically validated IHC assay
5. Barcelona Clinic Liver Cancer Stage B (if not amenable to local treatment/surgery) or C prior to apheresis
6. Child-Pugh score: Grade A
7. Participants with HBV and HCV undergoing management of these infections per institutional practice.

Exclusion Criteria:

1. Active or prior documented gastrointestinal (GI) variceal bleed or history of upper GI bleeding, ulcers, or esophageal varices with bleeding within 12 months
2. History of liver transplantation or on waiting list
3. Current clinically significant ascites
4. Main portal vein thrombus, or tumor thrombus invasion of mesenteric vein / inferior vena cava
5. Uncontrolled intercurrent illness
6. Active Infections
7. Positive serology for HIV
8. History of hepatic encephalopathy within 12 months prior to treatment allocation
9. History of chronic or recurrent (within the last year) severe autoimmune or immune mediated disease requiring steroids or other immune-suppressive treatments.
10. Prior treatment with any CAR-T therapy directed at any target or any therapy that is targeted to GPC3.
11. Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumour embolisation, or monoclonal antibodies, investigational product) within 5 half-lives or ≤ 21 days (whichever is shortest).

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2023-12-14 (Actual); Primary Completion 2027-12-13 (Estimated); Study Completion 2027-12-13 (Estimated)

PRIMARY OUTCOMES:
1. Incidence of participants with dose-limiting toxicities (DLTs), adverse events (AEs), including adverse events of special interest (AESI) and serious adverse events (SAEs). Determination of the recommended dose of AZD5851 for expansion phase | Through study completion, an average of 2 years
  Determine if treatment with AZD5851 is safe and tolerable through assessment of DLTs, AEs, SAEs and changes from baseline in vital signs, ECGs, and laboratory parameters

SECONDARY OUTCOMES:
1. Proportion of participants with a confirmed Complete Response (CR) or Partial Response (PR) | Through study completion, an average of 2 years
  Evaluation of the efficacy of the treatment by assessment of the Overall Response Rate according to RECIST v1.1 (ORR)
2. Interval between the date of AZD5851 infusion dose and first documented evidence of CR or PR | Through study completion, an average of 2 years
  Evaluation of the efficacy of the treatment by assessment of time to first response (TTR)
3. Proportion of participants who have a confirmed CR, PR, or who have stable disease (SD) for at least 5 weeks after the date of AZD5851 infusion | Through study completion, an average of 2 years
  Evaluation of the efficacy of the treatment by assessment of disease control rate according to RECIST v1.1 (DCR)
4. The proportion of participants who have a confirmed response (CR/PR) with a duration of at least a specific number of months | Through study completion, an average of 2 years
  Evaluation of the efficacy of the treatment by assessment of durable response rate according to RECIST v1.1 (DRR)
5. The best response the participant achieved according to RECIST v1.1 | Through study completion, an average of 2 years
  Evaluation of the efficacy of the treatment by assessment of best overall response according to RECIST v1.1 (BoR)
6. Interval between the date of first documented objective response date of first documented disease progression or the last evaluable assessment in the absence of progression | Through study completion, an average of 2 years
  Evaluation of the efficacy of the treatment by assessment of duration of response according to RECIST v1.1 (DoR)
7. Interval between the date of first T cell infusion and the earliest date of disease progression or death due to any cause | Through study completion, an average of 2 years
  Evaluation of the efficacy of the treatment by assessment of progression-free survival (PFS)
8. Interval between the date of first T cell infusion and date of death due to any cause | Through study completion, an average of 2 years
  Evaluation of the efficacy of the treatment by assessment of overall survival (OS)
9. Pharmacokinetics - maximum serum concentration of AZD5851 | Through study completion, an average of 2 years
  Maximum blood concentration (Cmax)
10. Pharmacokinetics -time to peak serum concentration of AZD5851 | Through study completion, an average of 2 years
  Time to peak (maximum) blood concentration (Tmax)
11. Pharmacokinetics -time to last measurable serum concentration of AZD5851 | Through study completion, an average of 2 years
  Time to last detectable blood concentration (Tlast)
12. Pharmacokinetics - Exposure of AZD5851 | Through study completion, an average of 2 years
  Area under the curve (AUC)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (15):
  - Research Site, Phoenix, Arizona
  - Research Site, Duarte, California
  - Research Site, Orange, California
  - Research Site, San Francisco, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Jacksonville, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Westwood, Kansas
  - Research Site, Rochester, Minnesota
  - Research Site, Hackensack, New Jersey
  - Research Site, New York, New York
  - Research Site, Columbus, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
- Japan (2):
  - Research Site, Kashiwa
  - Research Site, Osakasayama-shi
- Research Site, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/